CLINICAL TRIAL: NCT00000256
Title: Reinforcing Effects of Brief Exposures to Nitrous Oxide
Brief Title: Reinforcing Effects of Brief Exposures to Nitrous Oxide - 8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: NIDA-08391-8; R01DA008391 (NIH); R01-08391-8
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; reinforcer; subjective effects; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo + 20% N2O (Active Comparator): 0% N2O inhaled during psychomotor testing, 20% N2O inhaled during psycho motor testing, then subject's choice of the 2.
  Interventions: Drug: 20% N2O
- Placebo + 40% N2O (Active Comparator): 0% N2O inhaled during psychomotor testing, 40% N2O inhaled during psycho motor testing, then subject's choice of the 2.
  Interventions: Drug: 40% N2O
- Placebo + 60% N2O (Active Comparator): 0% N2O inhaled during psychomotor testing, 60% N2O inhaled during psycho motor testing, then subject's choice of the 2.
  Interventions: Drug: 60% N2O
- Placebo + 80% N2O (Active Comparator): 0% N2O inhaled during psychomotor testing, 80% N2O inhaled during psycho motor testing, then subject's choice of the 2.
  Interventions: Drug: 80% N2O

INTERVENTIONS:
Drug: 20% N2O
  Arms: Placebo + 20% N2O
Drug: 40% N2O
  Arms: Placebo + 40% N2O
Drug: 60% N2O
  Arms: Placebo + 60% N2O
Drug: 80% N2O
  Arms: Placebo + 80% N2O

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. Comparisons between nitrous oxide, opiates, and benzodiazepine antagonists will be made. To examine reinforcing effects of brief exposures to nitrous oxide in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Ages: 22 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 1995-08; Primary Completion 1996-11 (Actual); Study Completion 1996-11 (Actual)

PRIMARY OUTCOMES:
Choice of nitrous oxide vs placebo | After 1.5 min of inhalation each of nitrous oxide then placebo
  Subjects underwent 4 sessions consisting of 2 sample tests (inhaling placebo and inhaling varying doses of N2O), then choosing which inhalant they wanted for a choice test. The subject & the technician administering the inhalant were blinded. During each intervention and each session, subjects underwent psychomotor testing.

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Zacny JP, Klafta JM, Coalson DW, Marks S, Young CJ, Klock PA, Toledano AY, Jordan N, Apfelbaum JL. The reinforcing effects of brief exposures to nitrous oxide in healthy volunteers. Drug Alcohol Depend. 1996 Nov;42(3):197-200. doi: 10.1016/s0376-8716(96)01281-1. PMID 8912802